CLINICAL TRIAL: NCT01377545
Title: Continuous Infraclavicular Nerve Blocks: Needle Versus Catheter Local Anesthetic Bolus
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Associate Professor, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Infraclav Needle vs Catheter
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Nerve Block
Keywords: Infraclavicular; Nerve Block; Needle; Perineural Catheter; Volunteer; Upper Extremity Nerve Block; Sensation; Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local Anesthetic Via Catheter (Active Comparator): 30mL of Lidocaine (local Anesthetic) will be injected via a perineural catheter at hour 0.
  Interventions: Procedure: Local Anesthetic given via perineural catheter for infraclavicular nerve block.
- Local Anesthetic Via Needle (Active Comparator): 30mL of Lidocaine (local Anesthetic) will be injected via a needle at hour 0.
  Interventions: Procedure: Local Anesthetic given via needle for infraclavicular nerve block

INTERVENTIONS:
Procedure: Local Anesthetic given via perineural catheter for infraclavicular nerve block. — Patients will be randomized to receive 30mL of Lidocaine via Catheter for an infraclavicular nerve block on one side (right or left) and via needle on the other side. Sensory and strength will be tested following local anesthetic administration.
  Arms: Local Anesthetic Via Catheter
Procedure: Local Anesthetic given via needle for infraclavicular nerve block — Patients will be randomized to receive 30mL of Lidocaine via Catheter for an infraclavicular nerve block on one side (right or left) and via needle on the other side. Sensory and strength will be tested following local anesthetic administration.
  Arms: Local Anesthetic Via Needle

SUMMARY:
The investigators propose to test the hypothesis that when placing a perineural catheter for a continuous peripheral nerve block, injecting the initial local anesthetic bolus via the insertion needle results in a faster-onset sensory block than injecting the initial bolus via the perineural catheter. The study results will help define the optimal local anesthetic bolus introduction technique-needle versus catheter-for peripheral nerve blocks when placing a perineural catheter.

DETAILED DESCRIPTION:
Specific Aim: The investigators propose to test the hypothesis that when placing a perineural catheter for a continuous peripheral nerve block, injecting the initial local anesthetic bolus via the insertion needle results in a faster-onset sensory block than injecting the initial bolus via the perineural catheter. The study results will help define the optimal local anesthetic bolus introduction technique-needle versus catheter-for peripheral nerve blocks when placing a perineural catheter.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* willing to have bilateral infraclavicular blocks/catheters placed

Exclusion Criteria:

* current daily analgesic use
* opioid use within the previous 4 weeks
* any neuro-muscular deficit of either upper extremity
* body mass index > 30 kg/m2
* weight < 50 kg [100 lbs]
* pregnancy
* incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Sensory Level | 120 minutes
  EKG pads will be positioned in the 5 major nerve distributions distal to the elbow, ensuring placement is equivalent bilaterally. The primary endpoint will be the time, in minutes, until all 5 nerve territories record > 60 mA, or 120 minutes-whichever occurs first-since 60 mA is estimated to be equivalent to a surgical incision.

SECONDARY OUTCOMES:
Grip Strength | 120 Minutes
  Evaluated using a portable isometric force dynamometer to measure the maximum voluntary isometric contraction (MVIC) of the hand/fingers. Subjects will be asked to take 2 sec to come to maximum effort, maintain this effort for 3 sec, and then relax.
Sensory level for individual nerves | 120 Minutes
  Evaluated using transcutaneous electrical stimulation (TES) in the same manner as described for the primary end point.

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD CTRI, Hillcrest, San Diego, California, United States